CLINICAL TRIAL: NCT01485458
Title: Randomized Trial of Early Versus Delayed Surgery for Acute Traumatic Cervical Spinal Cord Injury Without Bone Injury in Patients With Cervical Canal Stenosis
Brief Title: Optimal Treatment for Spinal Cord Injury Associated With Cervical Canal Stenosis (OSCIS) Study
Acronym: OSCIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo University (Other)
Responsible Party: Principal Investigator, Hirotaka Chikuda, Lecturer, Tokyo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSCIS; UMIN000006780 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2011-11-30; First posted 2011-12-05 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Spinal Cord Injury
Keywords: Incomplete spinal cord injury; Cervical canal stenosis; Ossification of the posterior longitudinal ligament; Surgery; Decompression
MeSH Terms: conditions — Spinal Cord Injuries; Ossification of Posterior Longitudinal Ligament

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early surgery (Experimental)
  Interventions: Procedure: Early surgery
- Delayed surgery (Active Comparator)
  Interventions: Procedure: Delayed surgery

INTERVENTIONS:
Procedure: Early surgery — Surgery within 24 hours after admission
  Arms: Early surgery
Procedure: Delayed surgery — Surgery more than 2 weeks after injury
  Arms: Delayed surgery

SUMMARY:
Controversy exists regarding the optimal management of acute traumatic cervical spinal cord injury (SCI), especially those without bone injury. Although surgical decompression is often performed in SCI patients with cervical canal stenosis, efficacy and timing of surgery continues to be a subject of intense debate. In this randomized controlled trial, the investigators compare two strategies: early surgery within 24 hours after admission and delayed surgery following at least 2 weeks of conservative treatment. The purpose of this study is to examine whether early surgery would result in greater improvement in motor function as compared with delayed surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute traumatic cervical spinal cord injury (at C5 or below) admitted within 48 hours after injury

  1. No bone injury (no fracture or instability)
  2. American Spinal Injury Association (ASIA) Impairment Grade C
  3. Cervical canal stenosis due to preexisting conditions such as spondylosis and ossification of the posterior longitudinal ligament (OPLL)

Exclusion Criteria:

1. Unstable medical status
2. Difficult to undergo surgery within 24 hours after admission
3. Impaired consciousness or mental disorder that precludes neurological examination
4. Difficult to obtain informed consent in Japanese

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-12; Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
ASIA motor score | baseline and one year
  change from baseline to one year in the American Spinal Injury Association (ASIA) motor score
the ability to walk without assistance | one year
  proportion of patients who regained the ability to walk without assistance
Spinal Cord Independence Measure (SCIM) | one year
  the total score of the Spinal Cord Independence Measure (SCIM) version 3

SECONDARY OUTCOMES:
Health-related quality of life | one year
  SF-36 EQ-5D
Neuropathic pain | one year
  Neuropathic Pain Symptom Inventory
Walking status | one year
  Walking Index for Spinal Cord Injury (WISCI) II

CONTACTS AND LOCATIONS:
Overall Officials: Hirotaka Chikuda, MD, PhD, Principal Investigator — Tokyo University
Locations (1):
- The University of Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] OSCIS investigators; Chikuda H, Koyama Y, Matsubayashi Y, Ogata T, Ohtsu H, Sugita S, Sumitani M, Kadono Y, Miura T, Tanaka S, Akiyama T, Ando K, Anno M, Azuma S, Endo K, Endo T, Fujiyoshi T, Furuya T, Hayashi H, Higashikawa A, Hiyama A, Horii C, Iimoto S, Iizuka Y, Ikuma H, Imagama S, Inokuchi K, Inoue H, Inoue T, Ishii K, Ishii M, Ito T, Itoi A, Iwamoto K, Iwasaki M, Kaito T, Kato T, Katoh H, Kawaguchi Y, Kawano O, Kimura A, Kobayashi K, Koda M, Komatsu M, Kumagai G, Maeda T, Makino T, Mannoji C, Masuda K, Masuda K, Matsumoto K, Matsumoto M, Matsunaga S, Matsuyama Y, Mieda T, Miyoshi K, Mochida J, Moridaira H, Motegi H, Nakagawa Y, Nohara Y, Oae K, Ogawa S, Okazaki R, Okuda A, Onishi E, Ono A, Oshima M, Oshita Y, Saita K, Sasao Y, Sato K, Sawakami K, Seichi A, Seki S, Shigematsu H, Suda K, Takagi Y, Takahashi M, Takahashi R, Takasawa E, Takenaka S, Takeshita K, Takeshita Y, Tokioka T, Tokuhashi Y, Tonosu J, Uei H, Wada K, Watanabe M, Yahata T, Yamada K, Yasuda T, Yasui K, Yoshii T. Effect of Early vs Delayed Surgical Treatment on Motor Recovery in Incomplete Cervical Spinal Cord Injury With Preexisting Cervical Stenosis: A Randomized Clinical Trial. JAMA Netw Open. 2021 Nov 1;4(11):e2133604. doi: 10.1001/jamanetworkopen.2021.33604. PMID 34751757
- [Derived] Chikuda H, Ohtsu H, Ogata T, Sugita S, Sumitani M, Koyama Y, Matsumoto M, Toyama Y; OSCIS investigators. Optimal treatment for spinal cord injury associated with cervical canal stenosis (OSCIS): a study protocol for a randomized controlled trial comparing early versus delayed surgery. Trials. 2013 Aug 7;14:245. doi: 10.1186/1745-6215-14-245. PMID 23924165